CLINICAL TRIAL: NCT06239987
Title: The Effect of Care-oriented Practical Training on Nurses' Intensive and Critical Care Competence and Healthcare-associated Infection Indicators
Brief Title: The Effect of Care-oriented Practical Training on Nurses' Intensive and Critical Care Competency and HAIs Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Yeliz Karaçar, Research Assistant, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KAEK-800
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Intensive Care Unit; Health Care Associated Infection; Patient-Centered Care; Competence
Keywords: Intensive Care Nursing; Care-oriented Practical Training; Health Care Associated Infection; Intensive and Critical Care Nursing Competence
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: It is planned to give a care-oriented applied training program to intensive care nurses in groups of 13-15 people for 2 hours. The training content includes evidence-based practice recommendations for intensive and critical care, hand hygiene, hygiene practices in patients with special needs, and prevention and control of common HAIs. In the first stage of the training, practical training will be given by the intensive care coordinator and infection control nurse on the application model. In the second stage, patient care practices of a care team consisting of an intensive care nurse and care support staff will be observed. The training will be conducted interactively with narration, demonstration and question and answer techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care-oriented group (Experimental): Care-oriented practical training intervention is a 2-hour care-oriented applied group training program for intensive care nurses in groups of 13-15 people.
  Interventions: Behavioral: Care-oriented Practical Training

INTERVENTIONS:
Behavioral: Care-oriented Practical Training — The training content includes evidence-based practice recommendations for intensive and critical care, hand hygiene, hygiene practices in patients with special needs, and prevention and control of common HAIs. In the first stage of the training, practical training will be given by the intensive care coordinator and infection control nurse on the application model. In the second stage, patient care practices of a care team consisting of an intensive care nurse and care support staff will be observed. The training will be conducted interactively with narration, demonstration and question and answer techniques.

SUMMARY:
It was aimed to evaluate the effect of care-oriented practical training on the intensive and critical care competencies of nurses, the hand hygiene compliance rate of nurses and care support staff, and HAI indicators.

DETAILED DESCRIPTION:
Does care-oriented practical training increase nurses's intensive and critical care competencies? Does care-oriented practical training increase the hand hygiene compliance rate of nurses and care support staff? Does care-oriented practical training reduce HAI indicators in intensive care units?

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in the Adult Intensive Care Unit
* Working as a care support staff in an adult intensive care unit
* Volunteering to participate in research

Exclusion Criteria:

* Wanting to withdraw from the research
* Not being able to attend the final test (due to illness, leave, report, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Intensive and Critical Care Nursing Competence Scale | Before the Care Oriented Practical Training Intervention (October 2023) and one month after the training (November 2023)
  The mean score of Intensive and Critical Care Nursing Competence Scale
Nurse hand hygiene compliance | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention.
  Nurse hand hygiene compliance rate (%)
Care support staff hand hygiene compliance | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention.
  hand hygiene compliance rate (%) of care support staff
Central catheter-associated bloodstream infections | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Central catheter-associated bloodstream infections rate (%)
Ventilator-associated Event | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Ventilator-associated Event rate (%)
Catheter-associated Urinary Tract Infections | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Catheter-associated Urinary Tract Infections rate (%)

SECONDARY OUTCOMES:
Klebsiella spp. | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Klebsiella spp. n (%)
Enterococcus spp. | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Enterococcus spp.n (%)
Acinetobacter spp | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Acinetobacter spp. n (%)
Pseudomonas spp. | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Pseudomonas spp. n (%)
Enterobacterales | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Enterobacterales, n (%)
Candida | Health care-associated infection indicators in the intensive care unit 3 months before the Care-Oriented Practical Training Intervention and 3 months after the intervention
  Candida, n (%)

CONTACTS AND LOCATIONS:
Overall Officials: Şenay TAKMAK, Asst. Prof., Study Director — Kütahya Health Sciences University
Locations (1):
- Akdeniz University, Konyaalti, Antalya, Turkey (Türkiye)